CLINICAL TRIAL: NCT05470894
Title: APASL Post-COVID-19 Vaccination Liver Injury (APCOVLI Study)
Brief Title: Liver Injury After COVID-19 Vaccination
Status: Completed | Type: Observational
Sponsor: Humanity & Health Medical Group Limited (Other)
Collaborators: Tokyo University (Other); Nihon University School of Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: APCOVLI-2022-01
Record Dates: First submitted 2022-07-21; First posted 2022-07-22 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Subjects After COVID-19 Vaccination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COVID-19 Vaccination Group: Subjects who have received at lease one dose of approved COVID-19 vaccine
  Interventions: Biological: Approved COVID-19 vaccine

INTERVENTIONS:
Biological: Approved COVID-19 vaccine — Vaccination for COVI9-19

SUMMARY:
The COVID-19 pandemic, caused by the severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2), is still raging across the world and vaccination is expected to lead us out of this pandemic. Although the efficacy of these vaccines is beyond doubt, safety still remains a concern. Liver injury, such as autoimmune hepatitis (AIH), has been reported after COVID-19 vaccination. The aim of this prospective study is to investigate the spectrum and profile of liver injury after COVID-19 vaccination in Asia-Pacific region and to explore the potential risk factors for the development of liver injury.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have received at least one dose of approved COVID-19 vaccine;
* Volunteer to participate in this study.

Exclusion Criteria:

* No valid consent.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects after COVID-19 vaccination
Sampling Method: Non-Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Number of subjects with liver injury after COVID-19 vaccination | Within 24 weeks after COVID-19 vaccination
  The COVID-19 vaccine-related liver injury (such as elevated liver enzymes, total bilirubin, etc.) was recorded and its spectrum and profile were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: George Lau, MD, Principal Investigator — Humanity & Health Medical Group; Masao Omata, MD, PhD, Principal Investigator — Tokyo University; Tatsuo Kanda, MD, PhD, Principal Investigator — Nihon University School of Medicine
Locations (3):
- Humanity & Health Medical Group Limited, Hong Kong, Hong Kong
- Japan (2):
  - Nihon University School of Medicine, Tokyo
  - Tokyo University, Tokyo